CLINICAL TRIAL: NCT01263847
Title: The Effect of Galactooligosaccharide (GOS) Supplementation on Calcium Absorption and Retention in Female Adolescent Girls
Brief Title: Galactooligosaccharide (GOS) Supplementation and Calcium Absorption in Girls
Acronym: Friesland
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Friesland Foods (Unknown)
Responsible Party: Principal Investigator, Berdine Martin, Research Scientist, Nutrition Science, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Friesland
Record Dates: First submitted 2010-03-29; First posted 2010-12-21 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Osteoporosis
Keywords: Dietary Supplement: Galactooligosaccharide
MeSH Terms: conditions — Osteoporosis | interventions — 4'-galactooligosaccharide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- No Galactooligosaccharide (Placebo Comparator): 0 g galactooligosaccharide added to calcium-containing yogurt beverage
  Interventions: Dietary Supplement: Galactooligosaccharide
- 5 g Galactooligosaccharide (Active Comparator): 5 g galactooligosaccharide provided in two calcium-containing yogurt beverage (2.5 g in each drink) per day
  Interventions: Dietary Supplement: Galactooligosaccharide
- 10 g Galactooligosaccharide (Active Comparator): 10 g galactooligosaccharide added to two calcium-containing yogurt beverage (5 g in each drink) per day
  Interventions: Dietary Supplement: Galactooligosaccharide

INTERVENTIONS:
Dietary Supplement: Galactooligosaccharide — Zero, 5 or 10 g/day of galactooligosaccharide will be administered in two yogurt drinks containing about 300 mg total calcium each per day for three weeks. During a clinical visit following three weeks of consumption, zero, 2.5 or 5 g of galactooligosaccharide will be administered in the same yogurt with the addition of 15 mg Ca-44 (calcium chloride). Participants will be given one of the above yogurts at breakfast in addition to intravenously receiving 3.5 mg Ca-43 (calcium chloride) in 4 ml saline one hour after breakfast consumption.
  Other Names: Friesland

SUMMARY:
The purpose of this study is to determine the effects of galactooligosaccharide (GOS) supplementation on calcium absorption and and gut microbe profiles.

DETAILED DESCRIPTION:
Galactooligosaccharides (GOS) have been shown to have positive effects on calcium absorption in animals and postmenopausal women. This study aims to see whether the addition of fiber in the form of GOS to a calcium-containing yogurt drink will increase calcium absorption compared to placebo in a group of girls near menarche. Secondary outcomes are to assess physical fitness and determine the relationship between physical fitness and calcium absorption in adolescent girls as well as assess changes in gut microbiota. During this three phase, randomized, controlled crossover study, participants will consume yogurt drinks supplemented with 0, 2.5 or 5 grams of GOS twice daily for three weeks. Following each three week period, participants will complete a weekend clinical visit to measure calcium absorption. Height, weight, bone density and geometry, calcium absorption, gut microbiota and physical fitness will be measured. Effects of this GOS fiber intervention may help elucidate a mechanism of action for improving bone health with fiber supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Female between ages of 10 and 12
* Calcium intake of 900-1300 mg/d

Exclusion Criteria:

* Take medication that influences calcium metabolism
* Any disorder of calcium or bone homeostasis
* BMI>90th percentile for age
* Smoking, illegal drug consumption
* Any gastrointestinal disease (crohn's disease, celiac disease, inflammatory bowel disease)
* Any disease affecting kidney function
* Broken bone within last 6 months
* Dislike of yogurt or yogurt drinks
* Regular use of foods containing probiotics or prebiotics

Ages: 10 Years to 12 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Calcium Absorption | baseline and 48 h urine and blood
  Calcium absorption will be measured using dual isotope methods. Calcium-44(Ca-44) as calcium chloride will be administered in a yogurt drink provided at breakfast along with a roll, butter, jam and juice. A second isotope, Calcium-43 (Ca-43) as calcium chloride will be administered intravenously, one hour after consumption of breakfast. Urine and blood samples will be collected over a period of 48 hours and levels of Ca-44 and Ca-43 will be measured in urine and blood. Levels of Ca-44 and Ca-43 will be expressed as a ratio (Ca-44/Ca-43).

SECONDARY OUTCOMES:
Change in fecal microbiota | after 3 weeks of product consumption

CONTACTS AND LOCATIONS:
Overall Officials: Connie M Weaver, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States